CLINICAL TRIAL: NCT01743846
Title: Accuracy of Continuous Non-invasive Arterial Pressure (CNAP) With Invasive Measurements Dependent on Cardiac Function, Vascular Resistance and Volume Status
Brief Title: CNAP Accuracy Dependent on Hemodynamic Variables
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, PD Dr. med Jochen Renner, University Hospital Schleswig-Holstein
Other Study IDs: CNAP 2010_3
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Accuracy and Precision of Noninvasive Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Major Surgery: Patients undergoing major surgery

SUMMARY:
Agreement of CNAP pressure with invasive pressure is evaluated dependent on hemodynamic variables achieved by a PICCO monitor.

Hypothesis: Low cardiac output and volume status but not high vascular resistance affect the accuracy of CNAP.

DETAILED DESCRIPTION:
Agreement of CNAP pressure with invasive pressure is evaluated dependent on hemodynamic variables achieved by a PICCO monitor.

Hypothesis: Low cardiac output and volume status but not high vascular resistance affect the accuracy of CNAP. Body mass index and age may have impact on the accuracy of PPV measured non-invasively on the basis of volume-clamp technique.

ELIGIBILITY:
Inclusion Criteria:

* need for invasive blood pressure measurement

Exclusion Criteria:

* age under 18
* emergencies
* cardiac dysrhythmia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major surgery under general anaesthesia
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
arterial pressure | intraoperative
  Accuracy and precision of CNAP in comparison with the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, PD Dr., Principal Investigator — University Hospital, Schleswig-Holstein. Departement of Anaesthesia and Intensive Care Medicine; Robert Hanss, Prof. Dr., Principal Investigator — University Hospital, Schleswig-Holstein. Departement of Anaesthesia and Intensive Care Medicine
Locations (1):
- University Hospital, Schleswig-Holstein. Departement of Anaesthesia and Intensive Care Medicine, Kiel, Germany